CLINICAL TRIAL: NCT06423638
Title: The Feasibility of Tai Chi Easy Training for Registered Nurses
Brief Title: Feasibility of Virtual Tai Chi Easy for Registered Nurses
Acronym: TCERN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Carlie Felion, PI, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003718
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Transition Shock; Nurses' Intention to Quit; Stress; Somatic Symptoms; Burnout; Trauma and Stressor Related Disorders
Keywords: Tai Chi Easy; Healthcare-Related Psychological Trauma; Virtual; Transition Shock; burnout; nurse; somatic symptoms; stress
MeSH Terms: conditions — Medically Unexplained Symptoms; Burnout, Psychological; Trauma and Stressor Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will complete two 60 minute virtual Tai Chi Easy classes per week and practice on their own 10 minutes per day on 4 other days each week for six weeks.
  Interventions: Behavioral: Virtual Tai Chi Easy

INTERVENTIONS:
Behavioral: Virtual Tai Chi Easy — The TCE intervention will be delivered asynchronously online. Participants can complete the classes at a time and in a location that is convenient for them. The classes will be offered for one hour twice weekly and were developed and recorded by a certified Tai Chi Easy practice leader.
  TCE is a simple form of mind-body self-care that focuses on four components:
  * Mindful movements that help to stretch, and relax the body while improving balance and coordination
  * Breathing practices that reduce stress by inducing a relaxation response while improving energy and circulation and enhancing innate healing responses
  * Self-applied massage to stimulate blood flow, relax the body, and improve circulation and energy
  * Meditation practices to relax the body, center the mind, and calm the emotions

SUMMARY:
This study will examine the feasibility of virtual Tai Chi Easy training for registered nurses and see if participation results in changes in symptoms of transition shock, healthcare-related psychological traumatic stress, burnout, somatic symptoms, and intention to quit. Participants will do virtual Tai Chi Easy for 2 hours per week and practice on their own for 40 minutes per week. The study will last six weeks. Surveys will be completed in REDCap before, during, and after the intervention.

DETAILED DESCRIPTION:
Nurses are the backbone of the healthcare system, comprising 59% of the healthcare workforce (Salmond, 2021); however, research indicates that 32.8% of newly hired Registered Nurses (RNs) voluntarily terminate their positions within the first year and must then be replaced (NSI Nursing Services, 2023). The turnover problem among nurses threatens the delivery of adequate, safe, and timely patient care, the health and well-being of nurses and other healthcare professionals, and the sustainability of the organizations for which they work.

High job turnover among nurses is a problem that has inspired the design, implementation, and study of numerous organization/system-driven interventions over at least the past sixty years. Numerous researchers have identified the first year of practice as the most stressful time in a nurse's career (Chesak, 2019), with the highest levels occurring at four and eight months of employment (Fang, 2022). These nurses can experience a phenomenon known as 'transition shock,' comprising cognitive, psychological, and emotional distress (Duchscher, 2009). Transition shock can lead to nurses feeling overwhelmed by the stark and unanticipated realities of nursing practice, especially if that reality conflicts with previously held ideals, beliefs, and expectations. In addition to experiencing elevated stress levels and transition shock, exposure to healthcare-related psychological trauma plays a key role in why nurses have left and continue to leave their positions and the profession in droves (Foli, 2019).

Burnout is a common phenomenon among nurses. Key contributors to the development of burnout among healthcare workers include exposure to traumatic events such as witnessing death and suffering, the psychological and physical demands of the job, shift work, low autonomy, inadequate social support, incivility in the workplace, low staffing, and poor communication and collaborative relationships with other healthcare professionals (Chesak, 2019).

Despite the significant human and financial resources invested in solutions that attempt to mitigate nurse turnover, there is surprisingly little evidence in the published literature on the use of integrative mind-body self-care interventions to help individual nurses cope with prolonged or toxic levels of stress, burnout, traumatic stress, and somatic symptoms.

Self-care deficits are common among nurses, who typically focus on helping and serving others. While altruism, compassion, and a commitment to help others draw many people to a career in nursing, the desire to help others deal with their health problems can sometimes overshadow a nurse's motivation or ability to care for themselves (Crane, 2016). A 2017 survey by the American Nurses Association (ANA, 2017) found that 68% of nurses put their patients' safety, health, and wellness ahead of their own. Furthermore, although nurses are well-educated and often teach patients about the importance of health-promoting behaviors, that knowledge does not always translate into engagement in healthy lifestyle behaviors among nurses themselves (Albert, 2014).

In the wake of the COVID-19 pandemic, when nurses are more traumatized, stressed, and spread thinner than ever (American Nurses Foundation, 2021), some are resorting to employing maladaptive coping strategies, such as substance or alcohol abuse, to cope with stress and negative emotions (Foli, 2021). This highly problematic engagement in maladaptive coping strategies highlights and underscores the need for safe, cost-effective, accessible, and acceptable self-care options for nurses.

Mind-body psychoneuroimmunology-based interventions, such as Tai Chi, have been used for centuries by people all over the world and may be a feasible self-care intervention for new graduate nurses. Mind-body therapies are defined as those that emphasize using the brain in conjunction with the body to harness innate healing powers. Mind-body exercise often includes multiple components, such as breathing practices, focused attention, meditation, and gentle physical movements (Bower, 2016). Numerous conceptual models propose that the primary mechanism by which mind-body therapies produce their effects is through self-regulation, which has a top-down effect on numerous physiological processes that impact health and health behaviors (Bower, 2016). Mind-body modalities can improve nurses' general health and well-being and may help prevent or reduce burnout by reducing psychological stress and alleviating somatic symptoms (Jung, 2021) through alterations in inflammatory processes (Irwin, 2015).

Tai Chi Easy™ (TCE) is a safe, cost-effective, non-pharmacological intervention developed by Dr. Roger Jahnke. TCE is a simplified and streamlined practice that draws from the four main recognized styles of tai chi (Ward, 2023). According to Jahnke (2003), the deliberate attention to breathing, movement, and meditation in tai chi integrates the nervous, endocrine, cardiovascular, digestive, and immune systems with the psyche.

TCE practice comprises four baskets: Self-applied massage, mindful movement, breathing exercises, and meditation exercises (Ward, 2023). TCE is appropriate for people of all ages and health conditions because it is easy to learn and perform and is extremely adaptable (Ward, 2023).TCE is a cost-effective and sustainable mind-body intervention that does not require any special clothing, footwear, or equipment and can be practiced virtually anywhere, at any time. Therefore, TCE is the ideal behavioral intervention for this study to help new nurses cope with stress and improve their overall health and well-being.

Offering TCE in an asynchronous, virtual format will allow nurses (who often work the night shift and may need to sleep when in-person classes would typically be offered) to allow for greater flexibility and opportunities to access the intervention.

The purpose of this study is to a) gain a deeper understanding of factors contributing to high turnover among nurses, including past exposure to adverse childhood experiences and adverse life events, b) determine whether virtual TCE training is a feasible, acceptable, safe, and appropriate mind-body self-care intervention among NGNs, and c) explore whether changes in stress, transition shock, posttraumatic stress symptoms, and transition shock occur after participation in a six-week asynchronous virtual TCE training intervention.

The specific aims of this study are as follows:

Aim 1: Feasibility

- Evaluate whether Tai Chi Easy™ is a feasible, acceptable, and appropriate self-care intervention for registered nurses. Recruitment, retention, intervention adherence, and safety data will also be obtained.

Aim 2: Changes in Symptoms of Distress

- Explore whether changes in stress, transition shock, burnout, somatic symptoms, posttraumatic stress symptoms, and intention to quit occur post-intervention.

The results of this study will 1) fill an important knowledge gap in the nursing literature, 2) inform future studies regarding the use of virtual Tai Chi Easy™ as a safe, acceptable, cost-effective, and sustainable intervention for nurses who may be experiencing the phenomena of interest, and 3) provide information with potential utility for the academic and healthcare industry sectors. There is a demonstrated need to better prepare nurses for the tumultuous and highly stressful entry to professional practice and to guide the design and implementation of programs to help new nurses adjust and remain in their roles.

ELIGIBILITY:
Inclusion Criteria:

Registered Nurses from any racial/ethnic, socioeconomic group, sex/gender. Access to a computer, tablet, or smartphone Reliable internet access Ability to read and write in English

Exclusion Criteria:

Refusal to provide informed consent Regularly participating in Tai Chi or other mind-body exercise (as defined by participating more than once per week) Refusal or inability to fully participate in the study protocol Previously diagnosed post-traumatic stress disorder not due to a healthcare-related exposure event, active substance use disorder, or serious mental illness.

An acute or chronic medical or mental health condition that would otherwise limit the person's ability to fully participate in study activities.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Virtual Tai Chi Easy training | 8 weeks
  Evaluating the feasibility, acceptability, and appropriateness of intervention, as well as recruitment and retention

SECONDARY OUTCOMES:
Transition Shock | 8 weeks
  Changes in characteristics of transition shock post-intervention
Burnout | 8 weeks
  Changes in burnout symptoms post intervention
Somatic Symptoms | 8 weeks
  Changes in somatic symptoms post intervention
Intention to Quit | 8 weeks
  Changes in intention to quit post-intervention
Stress and post-traumatic stress symptoms | 8 weeks
  Changes in stress and post-traumatic stress symptoms post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carlie M Felion, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers